CLINICAL TRIAL: NCT06712550
Title: Assessment of Maternal and Fetal Serum Soluble Fms-like Tyrosine Kinase-1, Seromucoid, and Protein-bound Hexose in Women With Pre-eclampsia: A Case-control Study
Brief Title: Assessment of Maternal and Fetal Serum Biomarkers in Women With Pre-eclampsia
Status: Completed | Type: Observational
Sponsor: SHAHLA KAREEM ALALAF (Other)
Responsible Party: Sponsor-Investigator, SHAHLA KAREEM ALALAF, Professor, Hawler Medical University
Organization: Hawler Medical University (Other)
Other Study IDs: HawlerMU6
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Markers; Preeclampsia Severe; Preeclampsia Mild; Umbilical Cord Issue; Inflammatory Response; Serum Seromucoid in Pregnancy; Protein-bound Hexose in Preeclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with Preeclampsia: This group will comprise pregnant women having preeclampsia who are scheduled to undergo either vaginal or cesarean delivery. Their blood and their newborn blood will be collected and tested for a panel of inflammatory markers. This research aims to explore the potential association between maternal and neonatal inflammatory profiles and the development of preeclampsia, as well as its impact on pregnancy outcomes. By examining these markers, we hope to gain a better understanding of the underlying inflammatory mechanisms involved in preeclampsia.
- Normotensive pregnant women: This group will consist of normotensive pregnant women during delivery who are scheduled to have their blood and their newborn blood tested for a panel of inflammatory markers and responses to inflammatory markers. One of the aims of this research is to investigate the potential association between maternal and neonatal inflammatory profiles in normotensive pregnancy in comparison to women with preeclampsia and their newborn By examining these markers

SUMMARY:
The findings of markers of placental dysfunction in women with preeclampsia may suggest that these biomarkers may be useful tools for early detection of preeclampsia

DETAILED DESCRIPTION:
Preeclampsia is a pregnancy-specific hypertension illness that is characterized by widespread maternal endothelial dysfunction and appears to be a systemic syndrome that originates in the placenta. Through binding to and blocking the interaction of placental growth factor (PlGF) and vascular endothelial growth factor (VEGF) with their receptors Flt1, soluble fms-like tyrosine kinase (sFlt1) functions as an antagonist of these growth factors. Most seromucoid and protein-bound hexose are released during an acute phase and are inflammatory glycoproteins. Hepatocytes in the liver, which are highly sensitive to stress, increase and leak into the bloodstream during any disease state. It is a time when the placenta demands more vascular development. In order to identify and explain the differences in sFLT-1, VEGF, PlGF levels, and inflammatory biomarker responses. Current study will investigate the differences in blood level of sFLT-1, VEGF, PLGF, Seromucoid and protein-bound hexose inflammatory biomarkers between those with PE (cases) and healthy pregnant women (controls).

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-45 years
* Gestational age of 26-41 weeks at the time of diagnosis for preeclampsia
* Delivered vaginally or abdominally
* Being of any parity (para 1 and more)
* Pregnancy being singleton or multiple pregnancies
* Willingness to provide informed consent

Exclusion Criteria:

* Pregnant woman having chronic hypertension
* Having Diabetes mellitus
* The lady on medications that can affect inflammatory markers or blood pressure
* Pregnant with fetal anomalies
* Refused to involve in the research

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: This case-control study will include 200 pregnant women(100 with preeclampsia and 100 normotensive). Umbilical cord blood samples will be collected from both groups at the time of delivery. Serum samples will be analyzed for a panel of inflammatory markers.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
To compare the levels of maternal and fetal serum soluble Fms-like tyrosine kinase-1 (sFlt-1), seromucoid, and protein-bound hexose between women with pre-eclampsia and a control group of healthy pregnant women. | one hour
  To quantify and compare the concentrations of soluble Fms-like tyrosine kinase-1 (sFlt-1), seromucoid, and protein-bound hexose in maternal and fetal serum between women diagnosed with pre-eclampsia and a control group of normotensive pregnant women.

SECONDARY OUTCOMES:
To assess the association between the levels of these biomarkers and the severity of pre-eclampsia. | one hour
  o quantify and compare the concentrations of soluble Fms-like tyrosine kinase-1 (sFlt-1), seromucoid, and protein-bound hexose in maternal and fetal serum between women diagnosed with pre-eclampsia and a control group of normotensive pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: SHAHLA K. ALALAF, prof., Study Director — Hawler Medical University; Jiyan L. Hussein, Assis. prof, Principal Investigator — Salahadin University, College of Science
Locations (1):
- Hawler Medical University, Erbil, Kurdistan Region, Iraq